CLINICAL TRIAL: NCT00704080
Title: A Phase 1 Dose-Escalation Study of XL765 (SAR245409) in Combination With Temozolomide With and Without Radiation in Subjects With Malignant Gliomas
Brief Title: A Study of XL765 (SAR245409) in Combination With Temozolomide With and Without Radiation in Adults With Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11441; XL765-002 (Other: (other study code))
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Mixed Gliomas; Malignant Gliomas; Glioblastoma Multiforme
Keywords: GBM; Anaplastic glioma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — XL765; Temozolomide

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL765 (SAR245409); Drug: Temozolomide

INTERVENTIONS:
Drug: XL765 (SAR245409) — Gelatin capsules supplied in 5-mg, 10-mg, and 50-mg strengths; continuous daily dosing
Drug: Temozolomide — Capsules supplied in 5-mg, 20-mg, 100-mg, 140-mg, 180-mg, and 250-mg strengths; dosed at 200 mg/m2/day for 5 consecutive days, repeated every 28 days
  Other Names: Temodar®

SUMMARY:
The purpose of this study is to determine the safety and tolerability of XL765 in combination with Temozolomide in adults with anaplastic gliomas or glioblastoma on a stable Temozolomide maintenance dose. XL765 is a new chemical entity that inhibits the kinases PI3K and mTOR. In preclinical studies, inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells, whereas inactivation of mTOR has been shown to inhibit the growth of tumor cells. Temozolomide (TMZ, Temodar®) is an orally administered alkylating agent with activity against malignant gliomas. It is approved by the Food and Drug Administration for the following indications: 1) treatment of newly diagnosed glioblastoma multiforme (GBM) patients when given concomitantly with radiotherapy and then as maintenance treatment; 2) refractory anaplastic astrocytoma (AA), ie, patients who have experienced disease progression on a drug regimen containing nitrosourea and procarbazine. Temozolomide is commonly used in the treatment of other anaplastic gliomas (AG) including oligodendroglial tumors and mixed gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intracranial Grade 3 or 4 anaplastic glioma or glioblastoma (astrocytic tumor, anaplastic oligodendroglioma, or oligoastrocytoma)
* Received prior standard radiation for a Grade 3 or 4 astrocytic tumor with a minimum cumulative dose of 40 Gy administered
* Completed at least one full cycle of temozolomide of 200 mg/m2/day administered on Days 1-5 of a 28-day cycle, without unacceptable toxicity or progression
* Karnofsky performance status of 60 or more
* Adequate organ and bone marrow function as defined by hematological and serum chemistry limits
* At least 18 years old.
* Both men and women must practice adequate contraception
* Informed consent

Exclusion Criteria:

* Progressed while on temozolomide
* Evidence of acute intracranial or intratumoral hemorrhage > Grade 1
* Restriction of some therapies/medications within specific timeframes prior to enrollment and during the study including cytotoxic chemotherapy other than temozolomide, biologic agents, nitrosoureas or mitomycin C, small-molecule kinase inhibitors, non-cytotoxic hormonal agents, prior therapy with a PI3K inhibitors, radiation therapy, enzyme-inducing anti-convulsants, valproic acid
* Not recovered from the toxic effects of prior therapy
* Pregnant or breast feeding
* History of diabetes mellitus
* Uncontrolled intercurrent illness
* Congestive heart failure, unstable angina, or a myocardial infarction within 3 months of entering the study.
* HIV positive
* Diagnosis of another malignancy may exclude subject from study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-08; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of XL765 administered in combination with temozolomide in subjects with anaplastic gliomas or glioblastoma currently stable on a maintenance temozolomide dose | Assessed at each visit/periodic visits

SECONDARY OUTCOMES:
To evaluate plasma pharmacokinetics and pharmacodynamic effects of XL765 and temozolomide when administered in combination | Assessed during periodic visits
To evaluate preliminary efficacy of XL765 in combination with temozolomide in adults with anaplastic gliomas or glioblastoma | Assessed during periodic visits

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (6):
  - Investigational Site Number, Birmingham, Alabama
  - Investigational Site Number, Los Angeles, California
  - Investigational Site Number, Boston, Massachusetts
  - Investigational Site Number, New York, New York
  - Investigational Site Number, Rochester, New York
  - Investigational Site Number, Cleveland, Ohio